CLINICAL TRIAL: NCT07056153
Title: Association Between Early Consultation by the Primary Care Physician After Hospitalization in Geriatric Medicine Department, and the Risk of Re-hospitalization at 1 and 3 Months
Acronym: GEREHOSP
Status: Recruiting | Type: Observational
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: GEREHOSP; 2025-A00157-42 (Other: ANSM)
Record Dates: First submitted 2025-06-27; First posted 2025-07-09 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Geriatric
Keywords: primary care physician; early post-hospitalization consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with consultation: Participation in this study includes a short telephone contact (5 to 10 minutes) at 1 and then at 3 months following discharge from hospital to answer several questions about the return home.
- Patient with no consultation: Participation in this study includes a short telephone contact (5 to 10 minutes) at 1 and then at 3 months following discharge from hospital to answer several questions about the return home.

SUMMARY:
The time it takes for patients to be readmitted to hospital is a major public health issue, both in terms of medical time and costs.

In fact, 15% of patients of all ages are likely to be re-hospitalized within a month of hospitalization.

Today, hospitalizations present a significant nosocomial risk, all the more so in fragile populations. If these hospitalizations are long or repeated, it is crucial to develop solutions to reduce their number.

Elderly people often have a number of complementary pathologies and frailties, which are frequently destabilized during hospitalization or on discharge.

In this context of medico-social and financial stakes, a 2012 survey showed that 86% of French physicians would be prepared to make themselves available within 24-48 hours of hospital discharge if the situation justified it. Changes in medical demographics are forcing primary care physicians to adapt their practices, and the evidence of a reduced risk of re-hospitalization would make it possible to prioritize the provision of this consultation on discharge from hospital.

Post-hospitalization follow-up consultations with the primary care physician are recommended, but investigators have very little data on their benefits.

Investigators hypothesise that an early consultation (1 month post-hospitalization at most) by an elderly patient's primary care physician after hospitalization in geriatric medicine promotes: patient follow-up; reduced risk of re-hospitalization within 3 months.

The aim of this study is to determine the association of an early consultation by the primary care physician in the month following discharge from geriatric medicine hospitalization with rehospitalization rates within 3 months.

DETAILED DESCRIPTION:
The time it takes for patients to be readmitted to hospital is a major public health issue, both in terms of medical time and costs. Indeed, 15% of patients of all ages are likely to be rehospitalized within a month of hospitalization.

From an economic point of view, in the United States in 2013, 20% of patients underwent an early rehospitalization, compared with around 15% in France in 2015, generating up to $26 billion in annual expenditure in the USA for these stays alone. Among the causes of these early rehospitalizations are cancer, heart, lung, liver and infectious diseases, most of which require close monitoring, especially for the most fragile populations.

Intrinsic risk factors such as age, the presence of multiple co-morbidities and a history of depression play an important role; but it has also been shown that extrinsic risk factors such as the presence or absence of therapeutic education, or re-hospitalizations for different medical reasons, are just as important. Another factor is the lack of access to primary resources (housing, food), to primary care (including primary care physician), pharmacies and transport. As a result, the risk of mortality within a year is three times higher than for patients who are not rehospitalized within less than 1 month.

Several studies estimate that 16% to 23% of re-hospitalizations within 30 days of discharge are avoidable. In this context, a number of programs have been proposed to reduce the rate of rehospitalization, particularly in patients with heart disease. For example, an interventional study showed that close follow-up over 3 months by an advanced practice nurse (APN) for patients initially hospitalized for myocardial infarction prolonged the time to the next readmission and reduced the number of deaths and, consequently, the cost of care. These parameters also improved with the intervention of an APN at the end of the hospital stay.

However, the populations studied in these interventional studies are very often patients with cardiac pathologies. Few of these studies look specifically at geriatric populations, even though the mean ages of the populations are very frequently over 60 years old. Focusing specifically on the elderly population, a systematic review in 2023 studying the risk factors for rehospitalization at 30 and 90 days, worldwide, found a risk of rehospitalization of 10.3% to 37.6% and 16% to 58% respectively.

Another systematic review, carried out in 2005 by the WHO, studied different types of hospital-city interaction: comprehensive geriatric assessment, discharge planning and therapeutic education. These interventions reduced re-hospitalization by 20% and early 6-month mortality in patients over 65 years old.

Furthermore, follow-up by a private nurse trained in geriatrics for 1 month, with a pre-established schedule, reduces the risk of readmission by around 17%, the risk of multiple readmissions by 12%, the length of hospital stay and, once again, the cost of care.

On the other hand, there is little data on the impact of early consultation by the primary care physician on discharge from hospital. This is all the more surprising given that a specific quotation for hospital discharge (MSH) was introduced in 2011 for the reasons given above, and its use is increasing year on year.

A general medicine thesis in 2020, studied the impact of ambulatory follow-up by the primary care physician, with an appointment scheduled within 7 days of hospitalization, prior to discharge from hospital, and observed a 10-fold reduction in the risk of readmission, all populations combined. Discharge to a care and rehabilitation unit is also a protective factor.

Another study, this time in the USA, showed that scheduling an appointment and systematically sending the report to the referring doctor before discharge from hospital reduced the readmission rate by 30%.

n this context of medico-social and financial stakes, a 2012 survey showed that 86% of French physicians would be prepared to make themselves available within 24-48 hours of hospital discharge if the situation justified it. Changes in medical demographics are forcing primary care physicians to adapt their practices, and the evidence of a reduced risk of re-hospitalization would make it possible to prioritize the provision of this consultation on discharge from hospital.

In this context, the aim of this descriptive observational study will be to determine the association of an early consultation by the primary care physician in the month following discharge from geriatric medicine hospitalization with rehospitalization rates within 3 months.

As the study is observational, it does not present any direct risks or benefits for patients, healthcare professionals or healthcare institutions.

If this study demonstrates the benefit of this early consultation, it could encourage primary care physician to carry out this consultation, thus potentially reducing mortality, nosocomial risk associated with multiple hospitalizations, and cost for society.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 75 years
2. Patients hospitalized in the geriatric department of one of the investigating centers
3. Patient discharged home from the geriatrics department of one of the investigating centers
4. No objection from patient or legal representative to participate in study

Exclusion Criteria:

1. Patients who do not have a primary care physician
2. Patients living in an institution or transferred to an institution

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥ 75 years, who were hospitalized in the geriatrics department of one of the 3 investigating centers
Sampling Method: Non-Probability Sample
Enrollment: 301 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Describe the impact of early consultation by the primary care physician in elderly patients who have been hospitalized in geriatric medicine. The early consultation must have taken place within one month of discharge. | At 1 month after the end of hospitalisation
  Rate of rehospitalization between initial hospital discharge and 3-month follow-up. This rehospitalization rate will be compared between the 2 groups (with and no consultation). At 1 month : date of consultation with the primary care physician, Number of unscheduled rehospitalizations.
Describe the impact of early consultation by the primary care physician in elderly patients who have been hospitalized in geriatric medicine. The early consultation must have taken place within one month of discharge. | At 3 months after the end of hospitalisation
  Rate of rehospitalization between initial hospital discharge and 3-month follow-up. This rehospitalization rate will be compared between the 2 groups (with and no consultation). At 3 months : date of consultation with the primary care physician, Number of unscheduled rehospitalizations.

SECONDARY OUTCOMES:
Demonstrate reduction in 1-month mortality | 1 month after the end of hospitalization
  1-month mortality
Demonstrate reduction in 3-month mortality | 3 month after the end of hospitalization
  3-month mortality
Demonstrate reduction in length of stay in hospital | At 3 month after the end of 1st hospitalization
  Number of days of unscheduled full hospitalization between discharge from 1st hospitalization and 3-month visit,
Demonstrate reduced care costs | At 3 months after the initial hospital admission
  Total cost of all care procedures between initial hospital admission and 3-month visit

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel EJ Jarry, Dr. general medicine, Principal Investigator — GHMG; Theo TV Ventura, project manager, Study Director — GHMG
Locations (3):
- France (3):
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble, Isere
  - Centre Hospitalier Universitaire Grenoble Alpes Site de Voiron, Voiron, Isere
  - Centre Hospitalier Métropole Savoie, Chambéry, Savoie

IPD SHARING:
Plan to Share IPD: No